CLINICAL TRIAL: NCT02473666
Title: Patient Blood Management - Use and Outcome
Acronym: PBM-USZ
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK 2015-0175
Record Dates: First submitted 2015-05-11; First posted 2015-06-16 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Hemorrhage
Keywords: Patient Blood Management; Red Blood Cells; Platelet
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Health Conditions.: All Health Conditions. Area of Focus: Transfusions of blood products.

SUMMARY:
Study the influence of transfusion related Patient Blood Management Program actions on transfusion-related outcome measures and cost.

DETAILED DESCRIPTION:
At the University Hospital of Zurich, an in-house designed monitoring and feedback system was introduced which electronically registers each transfusion of any allogeneic blood product, be it red blood cells, plasma or platelets as well as corresponding laboratory data. Results are reported quarterly to Department heads. The investigator analyzes whether the introduction of this monitoring and feedback system as part of a patient blood management Program has a significant influence on use of allogeneic blood product transfusions and transfusion-related costs, without compromising patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* Only case records, all discharged patients of the University Hospital of Zürich

Exclusion Criteria:

* Not discharged from our Hospital.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All cases of all in hospital patients. Area of Focus: Transfusions of blood products.
Sampling Method: Probability Sample
Enrollment: 250000 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Percentage of transfusions per participant | participants will be followed form date of hospital entry until date of discharge or date of death up to 3 years
  Participant wich had transfusion will be identified and the administrative, financial and clinical data will be compared to participants without transfusions

SECONDARY OUTCOMES:
Percentage of transfusion of any blood product per participant | participants will be followed form date of hospital entry until date of discharge or date of death up to 3 years
  Count of any blood products per case, QM Data
Cost of any blood product per participant | participants will be followed form date of hospital entry until date of discharge or date of death up to 3 years
  costs per case
Survey of Patient Blood Management System | participants will be followed form date of hospital entry until date of discharge or date of death up to 3 years
  clinical, financial,and administrative data of all participants will be reviewed on the focus on transfusions

CONTACTS AND LOCATIONS:
Overall Officials: Donat R Spahn, Prof, Principal Investigator — IFA University Hospital Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland